CLINICAL TRIAL: NCT00000139
Title: Herpetic Eye Disease Study (HEDS) II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NEI-38
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2009-09

CONDITIONS: Keratitis, Herpetic; Ocular Herpes Simplex; Herpes Simplex
Keywords: Herpes Simplex Stromal Keratitis
MeSH Terms: conditions — Keratitis, Herpetic; Herpes Simplex | interventions — Acyclovir

INTERVENTIONS:
Behavioral: Stress
Drug: Acyclovir

SUMMARY:
To determine whether early treatment (with oral acyclovir) of herpes simplex virus (HSV) ulcerations of the corneal epithelium prevents progression to the blinding complications of stromal keratitis and iridocyclitis.

To determine the efficacy of low-dose oral acyclovir in preventing recurrent HSV eye infection in patients with previous episodes of herpetic eye disease.

To determine the role of external factors (such as ultraviolet light or corneal trauma) and behavioral factors (such as life stress) on the induction of ocular recurrences of HSV eye infections and disease.

DETAILED DESCRIPTION:
Infection of the eye by herpes simplex virus (HSV) is a leading cause of corneal blindness in the United States and other countries. The infection can lead to corneal scarring and neovascularization, permanent endothelial dysfunction and corneal edema, secondary glaucoma, and cataract. Despite the availability of topical antiviral agents that are highly active against HSV keratitis, there is still no known effective method for reducing the frequency of recurrence or severity of stromal keratitis and iridocyclitis. In addition, the prognosis is poor for recovery of good vision following penetrating keratoplasty for actively inflamed or highly vascularized herpetic corneas.

On the basis of both animal and human studies, the antiviral agent acyclovir may both treat and prevent recurrence of HSV disease. However, no consensus yet exists on the use of acyclovir in the management and prevention of herpetic eye disease.

HEDS-II consists of two randomized, placebo-controlled trials that are assessing the role of oral acyclovir in the management of herpetic eye disease and one epidemiologic study that is investigating risk factors, including stress, for the development of ocular recurrences of the disease. The organizational structure consists of a national coordinating center, eight regional coordinating clinical centers, and approximately 60 clinical sites. The clinical sites where patients are enrolled and followed include both university-based and community-based practices.

Herpes Simplex Virus Epithelial Keratitis Trial: HEDS-EKT evaluated the benefit of oral acyclovir given during treatment of an acute HSV keratitis (dendritic or geographic keratitis) in preventing the occurrence of later blinding complications. Patients entered the trial within 7 days of onset. All patients received standard treatment with a topical antiviral and were randomized to receive either oral acyclovir (400 mg five times a day for 21 days) or a placebo. Patients had eight visits within a 12-month followup period. The primary outcome was the time to the first occurrence of stromal keratitis or iridocyclitis in the study eye (eye with epithelial keratitis at time of study entry). The HEDS-EKT recruitment goal was 502 patients.

Acyclovir Prevention Trial: HEDS-APT evaluated the benefit of long-term acyclovir treatment in patients with a recent history of HSV eye disease but no current active disease. To be eligible, a patient must have experienced any kind of ocular herpes simplex infection (blepharitis, conjunctivitis, keratitis, or iridocyclitis) in the preceding year. The infection must have been inactive and untreated for at least the previous 30 days. Patients were randomized to receive either oral acyclovir (400 mg twice a day) or placebo for 1 year. Five followup visits occurred during the 1-year treatment period and an additional three followup visits during the 6-month post-treatment period. Episodes of recurrent HSV eye disease during the trial were treated with topical corticosteroids and antivirals as indicated, but patients continued to receive the oral acyclovir or placebo for the entire 365-day period. The primary outcome was the time to the first recurrence of any type of HSV eye disease in either eye. The recruitment goal was 696 patients.

Ocular HSV Recurrence Factor Study: HEDS-RFS is evaluating the effect of psychological, environmental, and biological factors on recurrences of herpetic eye disease. Patients recruited into the HEDS-APT trial are eligible to participate in HEDS-RFS if they are 18 years or older. At entry, all subjects fill out a questionnaire to estimate the negative affectivity trait measure. Subjects also fill out a short questionnaire every week for 52 weeks to track acute and chronic stressors (e.g., illnesses, injuries, menstrual periods, sun exposure, emotional and financial stresses). The investigators ensure patient privacy by the patient's mailing of the weekly logs directly to the HEDS National Coordinating Center.

ELIGIBILITY:
Protocol-specific criteria are noted in the description above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1992-10

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Francis I. Proctor Foundation, University of California, San Francisco, San Francisco, California
  - Emory Eye Center, Atlanta, Georgia
  - Eye Center, University of Illinois, Chicago, Chicago, Illinois
  - Louisiana State University Eye Center, New Orleans, Louisiana
  - Department of Ophthalmology, The Mount Sinai Medical Center, New York, New York
  - Wills Eye Hospital, Cornea Clinic, Philadelphia, Pennsylvania
  - Cullen Eye Institute, Baylor College of Medicine, Houston, Texas
  - The Eye Institute, Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Dawson CR, Beck R, Wilhelmus KR, Cohen EJ. Herpetic eye disease study. You can help. Arch Ophthalmol. 1996 Jan;114(1):89-90. doi: 10.1001/archopht.1996.01100130085015. No abstract available. PMID 8540857
- [Background] A controlled trial of oral acyclovir for the prevention of stromal keratitis or iritis in patients with herpes simplex virus epithelial keratitis. The Epithelial Keratitis Trial. The Herpetic Eye Disease Study Group. Arch Ophthalmol. 1997 Jun;115(6):703-12. doi: 10.1001/archopht.1997.01100150705001. PMID 9194719
- [Background] Acyclovir for the prevention of recurrent herpes simplex virus eye disease. Herpetic Eye Disease Study Group. N Engl J Med. 1998 Jul 30;339(5):300-6. doi: 10.1056/NEJM199807303390503. PMID 9696640